CLINICAL TRIAL: NCT03802682
Title: A Randomized, Open-label, Two-way, Crossover Study to Evaluate the Relative Bioavailability of Apalutamide Administered Orally as Whole Tablets and as a Mixture in Applesauce in Healthy Subjects
Brief Title: A Study of Apalutamide Administered Orally as Whole Tablets and as a Mixture in Applesauce in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108562; 2018-003774-27 (EudraCT Number); 56021927PCR1024 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-01-11; First posted 2019-01-14 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — apalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Sequence AB (Experimental): Participants will receive a single dose of apalutamide 240 milligram (mg) (4*60 mg tablets) swallowed whole under fasted conditions on Day 1 of Treatment Period 1 (Treatment A [reference]) followed by a single dose of apalutamide 240 mg (4*60 mg tablets) as a dispersed mixture in applesauce under fasted conditions on Day 1 of Treatment Period 2 (Treatment B [test]). Study treatment periods will be separated by a washout interval of at least 42 days and no more than 56 days between doses.
  Interventions: Drug: Apalutamide
- Treatment Sequence BA (Experimental): Participants will receive a single dose of apalutamide 240 mg (4*60 mg tablets) as a dispersed mixture in applesauce under fasted conditions on Day 1 of Treatment Period 1 (Treatment B [test]) followed by a single dose of apalutamide 240 mg (4*60 mg tablets) swallowed whole under fasted conditions on Day 1 of Treatment Period 2 (Treatment A [reference]). Study treatment periods will be separated by a washout interval of at least 42 days and no more than 56 days between doses.
  Interventions: Drug: Apalutamide

INTERVENTIONS:
Drug: Apalutamide — Participants will receive apalutamide 240 mg as a whole tablets administered orally (Treatment A) or as a dispersed mixture in applesauce (Treatment B) under fasted condition.
  Other Names: JNJ-56021927 and ARN-509

SUMMARY:
The purpose of this study is to determine the bioavailability of apalutamide tablets administered orally as dispersed tablets mixed in applesauce relative to whole tablets under fasting conditions in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

* Must agree not to donate sperm for the purpose of reproduction during the study and for a minimum of 3 months after receiving the last dose of study drug
* Body mass index (BMI; weight [Kilogram{kg}/height^2 [meter {m}^2]) between 18 and 30 kg/m^2 (inclusive), and body weight not less than 50 kg
* Blood pressure (after the participant is sitting for at least 5 minutes) between 90 and 140 millimeters of Mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic. If blood pressure is out of range, up to 2 repeated assessments are permitted
* Nonsmoker within the last 2 months (calculated from the first dosing)
* A 12-lead Electrocardiogram (ECG) at screening consistent with normal cardiac conduction and function, including: (1) Sinus rhythm; (2) Pulse rate between 40 and 100 beats per minute (bpm); (3) QTc interval less than or equal to (<=) 450 milliseconds (ms) (corrected Fridericia; QTcF); (4) QRS interval of less than (<) 120 ms; (5) PR interval <210 ms; and (6) Morphology consistent with healthy cardiac conduction and function

Exclusion Criteria:

* Clinically significant abnormal values for hematology or clinical chemistry at screening or at admission to the study center as deemed appropriate by the investigator
* Clinically significant abnormal physical examination, vital signs, or 12 lead electrocardiogram (ECG) at screening or at admission to the study center as deemed appropriate by the investigator
* Has a history of significant multiple and/or severe allergies, or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food including to excipients of apalutamide or to apple or applesauce
* History of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for paracetamol, within 14 days before the first dose of the study drug is scheduled until completion of the study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | Day 1: Predose, 30 minutes, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose
  Cmax is the maximum observed plasma concentration.
Area Under the Plasma Concentration-time Curve From Time 0 to 72 hours (h) (AUC [0-72h] | Day 1: Predose, 30 minutes, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose
  AUC(0-72h) is area under plasma concentration-time curve from time zero to 72 hours.
Area Under the Plasma Concentration-time Curve From Time 0 to 168 hours (AUC[0-168h]) | Day 1: Predose, 30 minutes, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose
  AUC(0-168h) is area under plasma concentration-time curve from time zero to 168 hours.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Approximately 84 days
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- See also: A Randomized, Open-label, Two-way, Crossover Study to Evaluate the Relative Bioavailability of Apalutamide Administered Orally as Whole Tablets and as a Mixture in Applesauce in Healthy Subjects — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR108562&attachmentIdentifier=9e043bf8-0e10-4797-9adb-2079ca785ec7&fileName=REDACTED_56021927PCR1024_CSR_Synopsis.pdf&versionIdentifier=